CLINICAL TRIAL: NCT07393191
Title: Clinical Instrumental Evaluation of the Efficacy of a Cosmetic Product in Improving Skin Moisturization and Skin Barrier
Brief Title: Evaluation of Hydrating Cream Effect on Subjects With Dry Skin.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lacer S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IT0007726/24
Record Dates: First submitted 2026-01-14; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Dry Skin; Sensitive Skin; Cracked Skin

STUDY DESIGN:
Intervention Model Description: Subjects applied the product on one leg, while the other leg was used as control (without product application).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subjects applied tested product on one leg and the other leg was left untreated (control) (Experimental): Subjects applied tested product on right or left leg (as per randomization) and the other leg was left untreated and acted as control area. The product was applied twice a day during 1 month.
  Interventions: Other: Repairing cream
- Untreated (No Intervention): No product application

INTERVENTIONS:
Other: Repairing cream — The cream was applied twice a day for 1 month
  Arms: subjects applied tested product on one leg and the other leg was left untreated (control)

SUMMARY:
The goal of this clinical trial is to learn if a cosmetic product works to improve skin condition in adults with dry, very dry, sensitive and cracked skin showing discomfort. The main questions it aims to answer are:

* Does the cosmetic increase skin hydration and skin barrier function?
* Does the cosmetic improve skin discomfort signs? Researchers will compare the skin condition with and without product use to see if it works to improve dry, sensitive and cracked skin.

Participants will:

* Use cosmetic twice a day for 1 month
* Visit the research center on day 1, 2, 7 and 28 of product use for evaluations

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male subjects (without specific repartition)
* Caucasian ethnicity
* Aged between 18 and 65 years old
* Subjects with dry (<30 c.u.), very dry (<25 c.u.), sensitive and cracked skin
* Subjects must show all the listed skin discomforts (skin dryness, desquamation, skin tightness, and itching
* Subjects aware of the study procedures and having signed an informed consent form
* Subjects registered with National Health Service (NHS)
* Subjects certifying the truthfulness of the personal data disclosed to the investigator
* Subjects able to understand the language used in the investigation and to respect the instructions given by the investigator as well as able to respect the study constraints and specific requirements
* The pharmacological therapy (except for the pharmacological therapy in the non-inclusion criteria) should be stable for at least one month without any changes expected or planned during the study
* Commitment not to change the daily routine or the lifestyle
* Subject informed about the study procedures and having signed the privacy policy

Exclusion Criteria:

* Subjects who do not fit the inclusion criteria.
* Subjects with acute or chronic diseases able to interfere with the outcome of the study or that are considered dangerous for the subject or incompatible with the study requirements
* Subjects participating or planning to participate in other clinical trials
* Subjects deprived of freedom by administrative or legal decision or under guardianship
* Subjects not able to be contacted in case of emergency
* Subjects admitted to a health or social facility
* Subjects planning a hospitalization during the study
* Subjects who participated in a similar study without respecting an adequate washout period (14 days)
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications
* Cosmetic treatment known to interfere with the tested product (e.g.: laser, peeling)
* Subjects having a skin disease or condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* Subjects intolerant or allergic to one or more ingredients of the cosmetic product
* Subjects that have shown allergies or sensitivity to cosmetic products, drugs, patch or medical devices
* Subject breastfeeding, pregnant or not willing to take necessary precautions to avoid pregnancy during the study (for the women of childbearing potential)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Change in skin moisturization from baseline to 28 days | Change from baseline in skin hydration at 30min, 24 hours, 48 hours, 7 days and 28 days.
  Skin hydration defined as skin capacitance value measured by Corneometer. Higher value means more hydrated skin.
Change in skin barrier function from baseline to 28 days | Change from baseline in skin barrier function at 30min, 24 hours, 48 hours, 7 days and 28 days.
  Skin barrier function defined as transepidermal water loss value measured by Tewameter. Lower value means improved skin barrier function.

SECONDARY OUTCOMES:
Assessment of product acceptability | Subjects responded to questionnaires at 30min, 24 hours, 48 hours, 7 days and 28 days of product use.
  Subjects responded a questionnaire with questions regarding acceptability and subjective efficacy of the product. The outcome measurement was the % of the agreement with the question.

CONTACTS AND LOCATIONS:
Overall Officials: Enza Cestone, Principal Investigator — Complife
Locations (1):
- Complife Italia, San Martino Siccomario, Milano, Italy

IPD SHARING:
Plan to Share IPD: No
Only summary of the results to support the publication will be shared. No complete study documents will shared.

DOCUMENTS (1):
  • Study Protocol (2024-12-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT07393191/Prot_000.pdf